CLINICAL TRIAL: NCT00735488
Title: Summary of the Data From the Prevention Programme for Hemoglobinopathies in Northern Israel
Brief Title: Sickle Cell Anemia Screening and Prevention in Northern Israel
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Ministry of Health, Israel (Other Government)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0011-08-EMC
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Thalassemia; Sickle Cell Anemia
Keywords: Thalassemia; Sickle cell anemia; Carrier detection; Prenatal Diagnosis; Genetic counseling
MeSH Terms: conditions — Thalassemia; Anemia, Sickle Cell | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: Thalassemia Minor carriers
  Interventions: Other: Observational
- B: Sickle cell carriers
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Summary of data

SUMMARY:
Since 1987, a screening for β Thalassemia in pregnant women is carried on in northern Israel, and from 1999 all the samples were tested also for Hgb S, Hgb C, Hgb D, Hgb O Arab and others.

In this study, the investigators intend to summarize the results of this preventive program aiming to detect couples at risk for having offspring with Thalassemia or SCA, the compliance regard to genetic counseling and prenatal diagnosis and the incidence of new affected babies born.

ELIGIBILITY:
Inclusion Criteria: All pregnant women tested and their husband in those cases that the woman test revealed abnormal hemoglobin.

Exclusion Criteria: No exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The program for prevention of hemoglobinopathies in Northern Israel, instituted since 1987, covered the northern part of Israel, including the Jezreel valley, the Nazareth area, the upper Galilee, the Hula valley and the northern part of the seashore region7. The overall population in this region is about a million inhabitants with about 50 % of Arab population, and a significant percentage of them from Bedouin origin, a population that at least partially is of African origin.
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Number of carriers detected | End of study

SECONDARY OUTCOMES:
Couples referred for prenatal diagnosis | End of study

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Koren, MD, Principal Investigator — Pediatric Hematology Unit - Ha'Emek Medical Center - Afula - 18101 - Israel
Locations (1):
- Pediatric Hematology Unit - Ha'Emek Medical Center, Afula, Afula, Israel